CLINICAL TRIAL: NCT07021911
Title: Concomitant Radiotherapy and New Drugs in Metastatic Breast Cancer
Acronym: COMBaRT
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Sponsor
Other Study IDs: PAR 73.23 OSS
Record Dates: First submitted 2025-05-07; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer; Radiotherapy; Complications
Keywords: breast cancer; radiotherapy; stereotactic radiotherapy (SABR); side effects
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- ADC's group: Patients undergoing ADC's drugs such as Trastuzumab Emtansine (TDM1), Trastuzumab Deruxtecan, Sacituzumab Govitecan
  Interventions: Radiation: Radiotherapy
- Cyclin-dependent kinases 4 and 6 inhibitors (CDK4/6 group): Patients receiving Palbociclib or Ribociclib or Abemaciclib
  Interventions: Radiation: Radiotherapy
- Anti Human Epidermal Growth Factor Receptor 2 monoclonal antibodies (Anti-Her2 group): Patients receiving Trastuzumab or Trastuzumab Pertuzumab
  Interventions: Radiation: Radiotherapy
- IT group: Patients receiving Atezolizumab or Pembrolizumab
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Conventional fractionated radiotherapy, moderate hypofractionated radiotherapy, stereotactic radiotherapy (SABR)

SUMMARY:
The primary objective of the study is to describe the tolerance profile of radiation treatments performed during systemic treatment with new drugs (molecular targeted therapies, immunotherapy, others).

DETAILED DESCRIPTION:
Patients suffering from stage IV breast cancer undergoing a systemic treatment including: molecular targeted therapy, conjugated antibodies (ADCs), monoclonal antibodies, tyrosine kinase inhibitors (TKI), immunotherapy (ICIs), who are candidates for a radiation treatment (both palliative or curative), after being informed about the study and giving written informed consent, will be considered eligible for this observational study. This study aims to prospectively analyze the tolerance profile of radiation treatments performed during new generation systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from stage IV breast cancer
* Ongoing systemic treatment including: molecular targeted therapy, conjugated antibodies, monoclonal antibodies, tyrosine kinase inhibitors, immunotherapy (immunocheckpoint inhibitors)
* Candidates for radiation treatment (both palliative and curative).

Exclusion Criteria:

* Previous radiation treatment on the same site
* Absolute contraindications to radiotherapy
* Systemic treatment administered as part of a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from stage IV breast cancer undergoing systemic treatment including: molecular targeted therapy, conjugated antibodies, monoclonal antibodies, tyrosine kinase inhibitors, immunotherapy (immunocheckpoint inhibitors)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2029-05-17 (Estimated); Study Completion 2029-05-17 (Estimated)

PRIMARY OUTCOMES:
Toxicity of Radiotherapy Treatments | Baseline, at 3, 6 month, one year from the end of radiation treatment, then yearly up to 3 years
  Acute and Late Toxicity evaluated with CTCAE (Common Terminology Criteria for Adverse Events) scale v6.0

SECONDARY OUTCOMES:
Response to Radiotherapy treatments with curative intent | evaluated at 3 months, 6 months, 1 year from treatments
  Response classified according to RECIST (Response Evaluation Criteria in Solid Tumours) criteria
Pain response to Radiotherapy treatments with palliative intent | evaluated at 3 and 6 months after treatments
  Pain response classified according to NRS (Numering Pain Rating Scale); this scale ranges from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Higher scores correspond to worse outcomes.
Progression free survival (PFS) | every 3 months after radiation treatments
  assessed from the start of radiation treatment to progression, local recurrence, or death, whichever comes first.

CONTACTS AND LOCATIONS:
Locations (1):
- Radiation Oncology Department Fondazione Policlinico Campus BioMedico, Rome, Italy, Italy